CLINICAL TRIAL: NCT01709773
Title: Focal Ablation of High-grade Cervical Intraepithelial Neoplasia
Brief Title: Focal Ablation of Cervical Precancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12503
Record Dates: First submitted 2012-10-15; First posted 2012-10-18 (Estimated); Last update posted 2018-02-20 (Actual); Status verified 2018-02

CONDITIONS: High-grade Cervical Intraepithelial Neoplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Focal treatment arm (Experimental)
  Interventions: Procedure: Focal treatment

INTERVENTIONS:
Procedure: Focal treatment — Focal treatment of high-grade cervical intraepithelial neoplasia using laser ablation, cryotherapy, or loop electrosurgical excision procedure

SUMMARY:
This is a pilot cohort study of women undergoing focal ablation for high-grade cervical intraepithelial neoplasia (HGCIN). The cohort was recruited from the UCSF Dysplasia Clinics. The standard treatment involves treatment of the entire cervix. Women with HGCIN meeting inclusion criteria were recruited for enrollment into the pilot study of focal treatment. Upon enrollment, they underwent focal ablational treatment rather than standard ablational treatment of the cervix. Follow-up visits were conducted at 2 weeks and 6 months to assess safety, feasibility, and acceptability. The 6-month recurrence rate of HGCIN will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-45 yo
* Biopsy-confirmed high grade cervical intraepithelial neoplasia grade 2, 3, or 2/3
* Satisfactory colposcopy, i.e., the entire transformation zone is visible
* Lesion occupying <= 2 quadrants of the cervix.

Exclusion Criteria:

* Unsatisfactory colposcopy.
* Colposcopic lesion extending into the endocervical canal beyond colposcopic visualization.
* Endocervical curettage positive for high-grade cervical intraepithelial neoplasia.
* Suspicion for invasive cancer on colposcopic exam.
* Glandular dysplasia or atypical glandular cells on cytology.
* Unreliable for follow-up.
* Immunosuppression (HIV, transplant recipient, etc.)

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2013-01-17 (Actual); Primary Completion 2014-04-11 (Actual); Study Completion 2014-05-26 (Actual)

PRIMARY OUTCOMES:
Six-month recurrence rate of high-grade cervical intraepithelial neoplasia | six months

SECONDARY OUTCOMES:
Safety of focal treatment | six months
  Participants will be asked to report any adverse events following focal treatment. These events will be graded according to standard criteria (DAIDS).
Acceptability of focal treatment | six months
  Participants will be asked to respond to a survey at enrollment and follow-up asking whether they are satisfied with focal treatment as an alternative method of treatment.
Feasibility of focal treatment | enrollment
  Providers will be asked to provide information after each treatment regarding whether the treatment was technically feasible to perform.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Smith-McCune, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States